CLINICAL TRIAL: NCT01729754
Title: A 52-Week, Phase 3, Randomized, Active Comparator and Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety/Tolerability of Subcutaneous Tildrakizumab (SCH 900222/MK-3222), Followed by an Optional Long-Term Safety Extension Study, in Subjects With Moderate-to-Severe Chronic Plaque Psoriasis (Protocol No. MK-3222-011)
Brief Title: A Study to Evaluate the Efficacy and Safety/Tolerability of Subcutaneous Tildrakizumab (SCH 900222/MK-3222) in Participants With Moderate-to-Severe Chronic Plaque Psoriasis Followed by a Long-term Extension Study (MK-3222-011)
Acronym: reSURFACE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3222-011; 2012-001377-88 (EudraCT Number); P07771 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tildrakizumab 200 mg (Experimental): Participants receive tildrakizumab 200 mg subcutaneously (SC) on Weeks 0, 4, 16, 28, 40 and 52 and, optionally, every 12 weeks thereafter until Week 244, plus etanercept placebo (PBO) twice weekly until Week 12 and once weekly from Week 12 to Week 28.
  Interventions: Drug: Tildrakizumab 200 mg; Drug: Etanercept Placebo
- Tildrakizumab 100 mg (Experimental): Participants receive tildrakizumab 100 mg SC on Weeks 0, 4, 16, 28, 40 and 52 and, optionally, every 12 weeks thereafter until Week 244, plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
  Interventions: Drug: Tildrakizumab 100 mg; Drug: Etanercept Placebo
- Placebo (Placebo Comparator): Participants receive matching placebo to tildrakizumab SC on Weeks 0 and 4 plus etanercept placebo twice weekly up to Week 12 and once weekly from Week 12 to Week 28. Participants will be re-randomized 1:1 at Week 12 to receive tildrakizumab 200 mg or tildrakizumab 100 mg on Weeks 12, 16, 28, 40 and 52 and, optionally, every 12 weeks thereafter until Week 244.
  Interventions: Drug: Tildrakizumab Placebo; Drug: Etanercept Placebo
- Etanercept 50 mg (Active Comparator): Participants receive matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly up to Week 12 and once weekly from Week 12 to Week 28. Participants who don't achieve PASI-75, receive tildrakizumab 200 mg after Week 28 (Weeks 32, 36 and 48) and, optionally, every 12 weeks thereafter until Week 244.
  Interventions: Drug: Tildrakizumab Placebo; Drug: Etanercept 50 mg

INTERVENTIONS:
Drug: Tildrakizumab 200 mg — Tildrakizumab 200 mg administered SC. Each pre-filled syringe (PFS) or autoinjector (AI) contains 1 mL of solution, tildrakizumab 100 mg/mL.
  Other Names: SCH 900222, MK-3222
  Arms: Tildrakizumab 200 mg
Drug: Tildrakizumab 100 mg — Tildrakizumab 100 mg administered SC. Each PFS or AI contains 1 mL of solution, tildrakizumab 100 mg/mL.
  Other Names: SCH 900222, MK-3222
  Arms: Tildrakizumab 100 mg
Drug: Tildrakizumab Placebo — Matching placebo to tildrakizumab administered SC
  Arms: Etanercept 50 mg; Placebo
Drug: Etanercept Placebo — Matching placebo to etanercept administered SC
  Arms: Placebo; Tildrakizumab 100 mg; Tildrakizumab 200 mg
Drug: Etanercept 50 mg — Etanercept 50 mg administered SC
  Other Names: Embrel
  Arms: Etanercept 50 mg

SUMMARY:
This study is being conducted to evaluate the efficacy and safety/tolerability of tildrakizumab (SCH 900222/MK-3222) in a population of participants with moderate-to-severe plaque psoriasis. The primary hypotheses of the study are that tildrakizumab is superior to placebo in the treatment of moderate-to-severe chronic plaque psoriasis as measured by the proportion of participants achieving >= Psoriasis Area Sensitivity Index of 75% (PASI-75) response and the proportion of participants with a Physician's Global Assessment (PGA) score of "clear" or "minimal" with at least a 2 grade reduction from baseline at Week 12.

DETAILED DESCRIPTION:
The base study consists of a screening phase of up to 4 weeks followed by a treatment period of 52 weeks, and a 20-week follow-up period. The base study treatment period is divided into 3 sequential parts.

In Part 1 of the base study (Week 0 to Week 12), participants will be randomized to one of 4 study arms (Arm A: tildrakizumab 200 mg + matching placebo to etanercept; Arm B: tildrakizumab 100 mg + matching placebo to etanercept; Arm C: matching placebo to tildrakizumab + matching placebo to etanercept; Arm D: matching placebo to tildrakizumab + etanercept 50 mg).

In Part 2 of the base study (Week 12 to Week 28), participants in Arm A and Arm B will receive matching placebo to tildrakizumab to maintain blinding at Week 12 and will receive either tildrakizumab 200 mg (Arm A) or tildrakizumab 100 mg (Arm B) at Weeks 12 and 16. Participants in Arm A and Arm B will also receive matching placebo to etanercept once weekly through study Week 28. At study Week 12, Arm C participants will be re-randomized to receive their first dose of tildrakizumab 200 mg or tildrakizumab 100 mg, and will receive additional doses of study medication according to their re-randomized treatment assignment at Week 16. Participants in Arm C will also receive matching placebo to etanercept through treatment Week 28. Participants in Arm D will continue with once weekly doses of etanercept through study Week 28 in combination with matching placebo to tildrakizumab.

In Part 3 of the base study (Week 28 to Week 52), participants in Arm A with >= PASI-75 response at Week 28 will be re-randomized to either continue tildrakizumab 200 mg or receive tildrakizumab 100 mg at study Weeks 28, 40, and 52. Participants with >= PASI-50 response but < PASI-75 response will continue to receive tildrakizumab 200 mg every 12 weeks and those participants with < PASI-50 response will be discontinued from the study. Participants in Arm B with >= PASI-75 response at Week 28 will continue to receive tildrakizumab 100 mg every 12 weeks. Those with >= PASI-50 response but < PASI-75 response will be re-randomized to receive continued tildrakizumab 100 mg or tildrakizumab 200 mg every 12 weeks. Participants in Arm B with < PASI-50 response will be discontinued from the study. Participants in Arm C will continue to receive treatment every 12 weeks according to their re-randomized treatment assignment. Participants in Arm D that achieve >= PASI-75 response at Week 28 will be discontinued from the study. Those participants with < PASI-75 response at Week 28 will be crossed over to tildrakizumab 200 mg to receive doses at Weeks 32, 36 and 48.

Eligible participants that choose to enroll in the extension study will have an additional treatment period of up to 192 weeks and will be monitored for an additional 20 weeks in the follow-up period. Each participant will receive tildrakizumab 200 mg or tildrakizumab 100 mg every 12 weeks up to study Week 244 according to their treatment assignment at the conclusion of Part 3 of the base study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate-to-severe plaque psoriasis for at least 6 months prior to enrollment;
* Candidate for phototherapy or systemic therapy;
* Premenopausal female participants must agree to abstain from heterosexual activity or use a medically approved method of contraception or use appropriate effective contraception as per local regulations or guidelines
* For the extension study: must have completed Part 3 of the base study
* For the extension study: must have achieved at least a PASI-50 response by the end of Part 3 of the base study

Exclusion Criteria:

* Non-plaque forms of psoriasis
* Presence or history of severe psoriatic arthritis and is well-controlled on current treatment regimen
* Women of childbearing potential who are pregnant, intend to become pregnant, or are lactating
* Participant is expected to require topical therapy, phototherapy, or systemic therapy during the trial
* Presence of any infection or history of recurrent infection requiring treatment with systemic antibiotics
* Previous use of entanercept, tildrakizumab (MK-3222), or other interleukin-23 (IL-23)/T- helper cell 17 (Th-17) pathway inhibitors including p40, p19, and IL-17 antagonists
* Latex allergy or sensitivity
* Active or untreated latent tuberculosis (TB)
* For the extension study: women of child-bearing potential who are pregnant, intend to become pregnant within 6 months of completing the trial, or are breast feeding
* For the extension study: active or uncontrolled significant organ dysfunction or clinically significant laboratory abnormalities
* For the extension study: expected to require topical treatment, phototherapy, or systemic treatment during the extension study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2021-10-26 (Actual)

REFERENCES:
- [Result] Reich K, Papp KA, Blauvelt A, Tyring SK, Sinclair R, Thaci D, Nograles K, Mehta A, Cichanowitz N, Li Q, Liu K, La Rosa C, Green S, Kimball AB. Tildrakizumab versus placebo or etanercept for chronic plaque psoriasis (reSURFACE 1 and reSURFACE 2): results from two randomised controlled, phase 3 trials. Lancet. 2017 Jul 15;390(10091):276-288. doi: 10.1016/S0140-6736(17)31279-5. Epub 2017 Jun 6. PMID 28596043
- [Derived] Armstrong AW, Blauvelt A, Lebwohl M, Asahina A, Gogineni R, Griffiths CEM. Efficacy and safety of tildrakizumab in patients with early- vs. late-onset psoriasis. Br J Dermatol. 2025 Aug 18;193(3):442-450. doi: 10.1093/bjd/ljaf171. PMID 40365708
- [Derived] Thaci D, Gerdes S, Du Jardin KG, Perrot JL, Puig L. Efficacy of Tildrakizumab Across Different Body Weights in Moderate-to-Severe Psoriasis Over 5 Years: Pooled Analyses from the reSURFACE Pivotal Studies. Dermatol Ther (Heidelb). 2022 Oct;12(10):2325-2341. doi: 10.1007/s13555-022-00793-z. Epub 2022 Sep 13. PMID 36098877
- [Derived] Thaci D, Piaserico S, Warren RB, Gupta AK, Cantrell W, Draelos Z, Foley P, Igarashi A, Langley RG, Asahina A, Young M, Falques M, Pau-Charles I, Mendelsohn AM, Rozzo SJ, Reich K. Five-year efficacy and safety of tildrakizumab in patients with moderate-to-severe psoriasis who respond at week 28: pooled analyses of two randomized phase III clinical trials (reSURFACE 1 and reSURFACE 2). Br J Dermatol. 2021 Aug;185(2):323-334. doi: 10.1111/bjd.19866. Epub 2021 May 4. PMID 33544883
- [Derived] Kerbusch T, Li H, Wada R, Jauslin PM, Wenning L. Exposure-response characterisation of tildrakizumab in chronic plaque psoriasis: Pooled analysis of 3 randomised controlled trials. Br J Clin Pharmacol. 2020 Sep;86(9):1795-1806. doi: 10.1111/bcp.14280. Epub 2020 Mar 25. PMID 32162721
- [Derived] Elewski B, Menter A, Crowley J, Tyring S, Zhao Y, Lowry S, Rozzo S, Mendelsohn AM, Parno J, Gordon K. Sustained and continuously improved efficacy of tildrakizumab in patients with moderate-to-severe plaque psoriasis. J Dermatolog Treat. 2020 Dec;31(8):763-768. doi: 10.1080/09546634.2019.1640348. Epub 2019 Jul 22. PMID 31268369
- [Derived] Reich K, Warren RB, Iversen L, Puig L, Pau-Charles I, Igarashi A, Ohtsuki M, Falques M, Harmut M, Rozzo S, Lebwohl MG, Cantrell W, Blauvelt A, Thaci D. Long-term efficacy and safety of tildrakizumab for moderate-to-severe psoriasis: pooled analyses of two randomized phase III clinical trials (reSURFACE 1 and reSURFACE 2) through 148 weeks. Br J Dermatol. 2020 Mar;182(3):605-617. doi: 10.1111/bjd.18232. Epub 2019 Jul 18. PMID 31218661
- [Derived] Jauslin P, Kulkarni P, Li H, Vatakuti S, Hussain A, Wenning L, Kerbusch T. Population-Pharmacokinetic Modeling of Tildrakizumab (MK-3222), an Anti-Interleukin-23-p19 Monoclonal Antibody, in Healthy Volunteers and Subjects with Psoriasis. Clin Pharmacokinet. 2019 Aug;58(8):1059-1068. doi: 10.1007/s40262-019-00743-7. PMID 30915660

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The tables below present the Participant Flow for the Base Study only (Weeks 0 to 52: Part 1 for 12 weeks, Part 2 for 16 weeks, and Part 3 for 24 weeks).
Groups:
- Tildrakizumab 200 mg (Parts 1 & 2): Participants received tildrakizumab 200 mg subcutaneously (SC) on Weeks 0 and 4 (Part 1), and Week 16 (Part 2) plus etanercept placebo (PBO) twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 200 mg (Parts 1, 2, & 3): Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3): Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and tildrakizumab 100 mg SC on Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 100 mg (Parts 1 & 2): Participants received tildrakizumab 100 mg subcutaneously (SC) on Weeks 0 and 4 (Part 1), and Week 16 (Part 2) plus etanercept placebo (PBO) twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3): Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and tildrakizumab 200 mg SC on Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 100 mg (Parts 1, 2, & 3): Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Placebo (Part 1): Participants received PBO to tildrakizumab SC on Weeks 0 and 4 plus etanercept PBO twice weekly until Week 12 (Part 1).
- Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3): Participants received PBO to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 200 mg SC on Weeks 12 and 16 (Part 2) and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3): Participants received PBO to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 100 mg SC on Weeks 12 and 16 (Part 2) and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28
- Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3): Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly up to Week 12 and once weekly from Week 12 to Week 28. Participants who didn't achieve PASI-75 at Week 28, received tildrakizumab 200 mg SC at Weeks 32, 36 and 48.
Period: Part 1
Arm/Group | Tildrakizumab 200 mg (Parts 1 & 2) | Tildrakizumab 200 mg (Parts 1, 2, & 3) | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Tildrakizumab 100 mg (Parts 1, 2, & 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Started | 20 | 184 | 110 | 18 | 21 | 268 | 14 | 72 | 70 | 313
Completed | 6 | 184 | 110 | 6 | 21 | 268 | 0 | 72 | 70 | 289
Not Completed | 14 | 0 | 0 | 12 | 0 | 0 | 14 | 0 | 0 | 24
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 3
Not completed — Non-compliance with Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 7 | 0 | 0 | 5 | 0 | 0 | 6
Not completed — Other Protocol Specified Criteria | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Period: Part 2
Arm/Group | Tildrakizumab 200 mg (Parts 1 & 2) | Tildrakizumab 200 mg (Parts 1, 2, & 3) | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Tildrakizumab 100 mg (Parts 1, 2, & 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Started | 6 | 184 | 110 | 5 (1 participant completed Part 1 but did not enter Part 2) | 21 | 268 | 0 | 72 | 70 | 289
Completed | 0 | 184 | 110 | 0 | 21 | 268 | 0 | 69 | 66 | 277
Not Completed | 6 | 0 | 0 | 5 | 0 | 0 | 0 | 3 | 4 | 12
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 4
Not completed — Other Protocol Specified Criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 3
Arm/Group | Tildrakizumab 200 mg (Parts 1 & 2) | Tildrakizumab 200 mg (Parts 1, 2, & 3) | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Tildrakizumab 100 mg (Parts 1, 2, & 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Started | 0 | 170 (14 participants completed Part 2 but did not enter Part 3) | 110 | 0 | 21 | 237 (31 participants completed Part 2 but did not enter Part 3) | 0 | 69 | 66 | 121 (156 participants completed Part 2 but did not enter Part 3)
Completed | 0 | 165 | 105 | 0 | 17 | 224 | 0 | 66 | 65 | 114
Not Completed | 0 | 5 | 5 | 0 | 4 | 13 | 0 | 3 | 1 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Other Protocol Specified Criteria | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the study arms: Tildrakizumab 200 mg, Tildrakizumab 100 mg, Placebo, Etanercept 50 mg, as per the treatments administered in Part 1 (Baseline Period).
Groups:
- Tildrakizumab 200 mg (Part 1): Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 plus etanercept placebo twice weekly until Week 12 (Part 1).
- Tildrakizumab 100 mg (Part 1): Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 plus etanercept placebo twice weekly until Week 12 (Part 1).
- Placebo (Part 1): Participants received tildrakizumab placebo SC at Weeks 0 and 4 and etanercept placebo SC twice weekly until Week 12 (Part 1).
- Etanercept 50 mg (Part 1): Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly until Week 12.
- Total: Total of all reporting groups
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1) | Etanercept 50 mg (Part 1) | Total
Number analyzed (Participants) | 314 | 307 | 156 | 313 | 1090
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (13.62) | 44.6 (13.59) | 46.4 (12.20) | 45.8 (13.97) | 45.2 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 87 | 44 | 91 | 311
  Male | 225 | 220 | 112 | 222 | 779
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 14 | 9 | 3 | 10 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 8 | 7 | 1 | 8 | 24
  White | 284 | 279 | 144 | 289 | 996
  More than one race | 2 | 7 | 3 | 3 | 15
  Unknown or Not Reported | 6 | 4 | 4 | 2 | 16
Body weight [Count of Participants; unit: Participants]
  <=90 kg | 180 | 176 | 90 | 180 | 626
  >90 kg | 134 | 131 | 66 | 133 | 464
Prior exposure to biologic therapy for psoriasis [Count of Participants; unit: Participants] — The following therapies constitute biologics therapy for psoriasis: efalizumab (RAPTIVA®), alefacept (AMEVIVE®), infliximab (REMICADE®), adalimumab (HUMIRA®), ustekinumab (STELARA®), and etanercept (Enbrel®)
  Participants
    Yes | 38 | 39 | 20 | 37 | 134
    No | 276 | 268 | 136 | 276 | 956
Psoriasis Area Sensitivity Index (PASI) [Mean (Standard Deviation); unit: Score on a scale] — The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. Population: Analysis populations includes randomized participants with PASI value at baseline.
  Score on a scale
    number analyzed (Participants) | 314 | 307 | 155 | 312 | 1088
    (all) | 19.8 (7.52) | 20.5 (7.63) | 20.0 (7.57) | 20.2 (7.36) | 20.1 (7.51)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Psoriasis Area Sensitivity Index 75% (PASI-75) Response at Week 12 (Part 1)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-75 response indicates the number of participants achieving a 75% reduction in PASI score compared to baseline. Statistical analyses presented below compare tildrakizumab to placebo to support the primary hypothesis of the study.
Time Frame: Week 12
Population: Analysis population includes all randomized participants who received at least 1 dose of Part 1 study treatment based on the treatment assigned.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 200 mg: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 plus etanercept placebo twice weekly until Week 12.
- Tildrakizumab 100 mg: Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 plus etanercept placebo twice weekly until Week 12.
- Placebo: Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 plus etanercept placebo twice weekly until Week 12.
- Etanercept 50 mg: Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly until Week 12.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Percentage of participants | 65.6 | 61.2 | 5.8 | 48.2
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (<=90kg, >90kg) and prior exposure to biologic therapy for psoriasis (yes/no). P-values are not adjusted for multiplicity; Difference in percentages = 59.8, 95% CI 2-sided [52.9 to 65.9] — Difference and confidence intervals (CIs) are calculated using Miettinen-Nurminen stratified by body weight (<=90kg, >90kg) and prior exposure to biologic therapy for psoriasis (yes/no) with sample size weights
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 55.5, 95% CI 2-sided [48.3 to 61.8] — Difference and CIs are calculated using Miettinen-Nurminen stratified by body weight (<=90kg, >90kg) and prior exposure to biologic therapy for psoriasis (yes/no) with sample size weights

2. Primary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 12 (Part 1)
Description: The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5. Statistical analyses presented below compare tildrakizumab to placebo to support the primary hypothesis of the study.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Percentage of participants | 59.2 | 54.7 | 4.5 | 47.6
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 54.7, 95% CI 2-sided [47.9 to 60.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Stratified by body weight (<=90kg, >90kg) and prior exposure to biologic therapy for psoriasis (yes/no). P-values are not adjusted for multiplicity; Difference in percentages = 50.2, 95% CI 2-sided [43.2 to 56.5] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) Up to Week 12 (Part 1)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 12
Population: Analysis population includes participants who took at least one dose of Part 1 study drug based on the treatment actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Percentage of participants | 49.4 | 44.3 | 55.1 | 54.0

4. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE Up to Week 12 (Part 1)
Description: as for outcome 3
Time Frame: Up to Week 12
Population: Analysis population includes participants who took at least one dose of Part 1 study medication based on the treatment actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Percentage of participants | 1.0 | 1.0 | 1.3 | 1.9

5. Secondary Outcome: Percentage of Participants Achieving a PASI-75 Response at Week 28 (Part 2)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-75 response indicates the number of participants achieving a 75% reduction in PASI score compared to baseline. Primary analysis for this endpoint is for participants randomized to tildrakizumab 200 mg, tildrakizumab 100 mg, or etanercept in Part 1.
Time Frame: Week 28
Population: Analysis population includes all participants randomized to tildrakizumab or etanercept in Part 1 who received at least one dose of study medication in Part 2.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 200 mg: Participants received tildrakizumab 200 mg SC on Weeks 0, 4, 16, and 28 plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 100 mg: Participants received tildrakizumab 100 mg SC on Weeks 0, 4, 16, and 28 plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Etanercept 50 mg: Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly up to Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 299 | 294 | 289
Percentage of participants | 72.6 | 73.5 | 53.6
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]; Difference in percentages = 19.2, 95% CI 2-sided [11.5 to 26.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]; Difference in percentages = 20.1, 95% CI 2-sided [12.4 to 27.6] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Achieving a PASI-75 Response at Week 40 (Part 3)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-75 response indicates the number of participants achieving a 75% reduction in PASI score compared to baseline. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Week 40
Population: Participants who received at least one dose of study medication in Part 3 and with valid PASI value at baseline and at Week 40.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 200 mg in Part 1 who were PASI responders at Week 28.
- Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and tildrakizumab 100 mg SC on Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 200 mg in Part 1 who were PASI responders at Week 28 and re-randomized to tildrakizumab 100 mg at Week 28.
- Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R: Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 100 mg in Part 1 who were PASI responders at Week 28.
- Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 200 mg in Part 1 who were PASI partial responders at Week 28.
- Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR: Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and tildrakizumab 200 mg SC on Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 100 mg in Part 1 who were PASI partial responders at Week 28 and re-randomized to tildrakizumab 200 mg at Week 28.
- Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR: Participants received tildrakizumab 100 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 100 mg in Part 1 who were PASI partial responders at Week 28.
- Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3): Participants received PBO to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 200 mg SC on Weeks 12 and 16 (Part 2) and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants who were randomized to placebo in Part 1 and who were re-randomized to tildrakizumab 200 mg for Part 2.
- Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3): Participants received PBO to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 100 mg SC on Weeks 12 and 16 (Part 2) and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants who were randomized to placebo in Part 1 and who were re-randomized to tildrakizumab 100 mg for Part 2.
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 107 | 108 | 212 | 60 | 21 | 21 | 67 | 64 | 114
Percentage of participants | 96.3 | 92.6 | 97.6 | 63.3 | 66.7 | 61.9 | 82.1 | 68.8 | 57.0

7. Secondary Outcome: Percentage of Participants Achieving a PASI-75 Response at Week 52 (Part 3)
Description: as for outcome 6
Time Frame: Week 52
Population: Participants who received at least one dose of study medication in Part 3 and with valid PASI value at baseline and at Week 52.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28, 40 and 52 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28. Arm includes participants randomized to tildrakizumab 200 mg in Part 1 who were PASI responders at Week 28.
- Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3): Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4 and etanercept 50 mg twice weekly up to Week 12 and once weekly from Week 12 to Week 28. Participants who didn't achieve PASI-75 at Week 28, received tildrakizumab 200 mg SC at Weeks 32, 36 and 48. Arm includes participants who were non-responders or partial responders to etanercept and re-randomized at Week 28 to receive tildrakizumab 200 mg.
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 104 | 204 | 60 | 19 | 19 | 66 | 63 | 113
Percentage of participants | 97.1 | 94.2 | 93.6 | 66.7 | 78.9 | 68.4 | 92.4 | 85.7 | 81.4

8. Secondary Outcome: Percentage of Participants With a PGA Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 28 (Part 2)
Description: The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5.
Time Frame: Week 28
Population: Analysis population includes participants randomized to tildrakizumab 100 mg, tildrakizumab 200 mg, or etanercept in Part 1 who received at least one dose of study medication in Part 2.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 100 mg: Participants received tildrakizumab 100 mg SC on Weeks 0, 4, 16 and 28 plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 299 | 294 | 289
Percentage of participants | 69.2 | 64.6 | 45.3
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 24.1, 95% CI 2-sided [16.2 to 31.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 19.6, 95% CI 2-sided [11.7 to 27.3] — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Percentage of Participants With a PGA Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 40 (Part 3)
Description: The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Week 40
Population: Participants who received at least one dose of study medication in Part 3 and with valid PGA value at baseline and at Week 40.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 107 | 106 | 212 | 59 | 21 | 21 | 66 | 64 | 112
Percentage of participants | 83.2 | 79.2 | 84.9 | 57.6 | 38.1 | 57.1 | 75.8 | 62.5 | 50.9

10. Secondary Outcome: Percentage of Participants With a PGA Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 52 (Part 3)
Description: as for outcome 9
Time Frame: Week 52
Population: Participants who received at least one dose of study medication in Part 3 and with valid PGA value at baseline and at Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 103 | 204 | 59 | 19 | 19 | 66 | 63 | 111
Percentage of participants | 84.8 | 77.7 | 79.4 | 50.8 | 42.1 | 57.9 | 77.3 | 55.6 | 68.5

11. Secondary Outcome: Percentage of Participants Achieving a PASI-90 Response at Week 12 (Part 1)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-90 response indicates the number of participants achieving a 90% reduction in PASI score compared to baseline.
Time Frame: Week 12
Population: Analysis population includes randomized participants who received at least one dose of study medication in study Part 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Percentage of participants | 36.6 | 38.8 | 1.3 | 21.4
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 35.3, 95% CI 2-sided [29.2 to 41.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 37.5, 95% CI 2-sided [31.1 to 43.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 15.2, 95% CI 2-sided [8.3 to 22.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 17.4, 95% CI 2-sided [10.3 to 24.4] — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Percentage of Participants Achieving a PASI-90 Response at Week 28 (Part 2)
Description: as for outcome 11
Time Frame: Week 28
Population: Analysis population includes participants randomized to tildrakizumab 100 mg, tildrakizumab 200 mg, or etanercept in Part 1 who received at least one dose of study medication in study Part 2.
Measure: Number; unit: Percentage of participants
Groups:
- Tildrakizumab 100 mg: Participants received tildrakizumab 100 mg SC on Weeks 0, 4 and 16 plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 293 | 290 | 277
Percentage of participants | 57.7 | 55.5 | 30.7
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]; Difference in percentages = 27.1, 95% CI 2-sided [19.1 to 34.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 24.9, 95% CI 2-sided [17.0 to 32.6] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Percentage of Participants Achieving a PASI-90 Response at Week 40 (Part 3)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-90 response indicates the number of participants achieving a 90% reduction in PASI score compared to baseline. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Week 40
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 107 | 108 | 212 | 60 | 21 | 21 | 67 | 64 | 114
Percentage of participants | 76.6 | 73.1 | 78.8 | 28.3 | 23.8 | 42.9 | 64.2 | 48.4 | 24.6

14. Secondary Outcome: Percentage of Participants Achieving a PASI-90 Response at Week 52 (Part 3)
Description: as for outcome 13
Time Frame: Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 104 | 204 | 60 | 19 | 19 | 66 | 63 | 113
Percentage of participants | 81.9 | 68.3 | 78.4 | 31.7 | 26.3 | 42.1 | 63.6 | 47.6 | 41.6

15. Secondary Outcome: Percentage of Participants Achieving a PASI-100 Response at Week 12 (Part 1)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-100 response indicates the number of participants achieving a 100% reduction in PASI score compared to baseline.
Time Frame: Week 12
Population: Analysis population includes randomized participants who received at least one dose of study medication in study Part 1 and with valid PASI value at baseline and Week 12.
Measure: Number; unit: Perentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 156 | 313
Perentage of participants | 11.8 | 12.4 | 0 | 4.8
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 11.7, 95% CI 2-sided [7.8 to 16.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 12.4, 95% CI 2-sided [8.5 to 16.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 7.0, 95% CI 2-sided [2.8 to 11.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 7.6, 95% CI 2-sided [3.3 to 12.3] — [estimate comment as in outcome 1, analysis 2]

16. Secondary Outcome: Percentage of Participants Achieving a PASI-100 Response at Week 28 (Part 2)
Description: as for outcome 15
Time Frame: Week 28
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 293 | 290 | 277
Percentage of participants | 27.0 | 22.8 | 11.2
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 15.7, 95% CI 2-sided [9.4 to 22.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 11.7, 95% CI 2-sided [5.6 to 17.9] — [estimate comment as in outcome 1, analysis 2]

17. Secondary Outcome: Percentage of Participants Achieving a PASI-100 Response at Week 40 (Part 3)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-100 response indicates the number of participants achieving a 100% reduction in PASI score compared to baseline. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Week 40
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 107 | 108 | 212 | 60 | 21 | 21 | 67 | 64 | 114
Percentage of participants | 39.3 | 38.9 | 33.5 | 11.7 | 0 | 14.3 | 29.9 | 28.1 | 5.3

18. Secondary Outcome: Percentage of Participants Achieving a PASI-100 Response at Week 52 (Part 3)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-100 response indicates the number of participants achieving a 90% reduction in PASI score compared to baseline. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 104 | 204 | 60 | 19 | 19 | 66 | 63 | 113
Percentage of participants | 46.7 | 37.5 | 35.3 | 10.0 | 5.3 | 31.6 | 39.4 | 23.8 | 15.9

19. Secondary Outcome: Baseline Dermatology Life Quality Index (DLQI)
Description: The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Time Frame: Baseline
Population: Analysis population includes randomized participants who received at least one dose of study medication with baseline and post-baseline DLQI values in Part 1.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 312 | 307 | 156 | 312
Score on a scale | 13.2 (7.03) | 14.8 (7.24) | 13.7 (6.98) | 14.5 (7.20)

20. Secondary Outcome: Change From Baseline in the DLQI at Week 12 (Part 1)
Description: as for outcome 19
Time Frame: Baseline and Week 12
Population: Analysis population includes randomized participants who received at least one dose of study medication with baseline or post-baseline DLQI values in Part 1.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 312 | 307 | 156 | 312
Score on a scale | -10.3 [-11.0 to -9.7] | -10.2 [-10.9 to -9.6] | -2.0 [-2.9 to -1.1] | -8.9 [-9.6 to -8.3]
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Other; p < 0.001, cLDA; Terms for time, the interaction of time by treatment, body weight (<=90 kg, >90 kg), and prior exposure to biologic therapy for psoriasis (yes/no); Difference in least squares means = -8.2, 95% CI 2-sided [-9.3 to -7.2]
Statistical Analysis 2: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Other; p < 0.001, cLDA; [statistical method as in outcome 20, analysis 1]; Difference in least squares means = -8.3, 95% CI 2-sided [-9.3 to -7.3]
Statistical Analysis 3: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Other; p = 0.002, cLDA; [statistical method as in outcome 20, analysis 1]; Difference in least squares means = -1.3, 95% CI 2-sided [-2.1 to -0.5]
Statistical Analysis 4: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Other; p = 0.001, cLDA; [statistical method as in outcome 20, analysis 1]; Difference in least squares means = -1.4, 95% CI 2-sided [-2.2 to -0.6]

21. Secondary Outcome: Change From Baseline in the DLQI at Week 28 (Part 2)
Description: as for outcome 19
Time Frame: Baseline and Week 28
Population: Analysis population includes randomized participants who received at least one dose of study medication and with baseline or post-baseline DLQI values in Part 1 or Part 2.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Tildrakizumab 100 mg: Participants received tildrakizumab 100 mg SC on Weeks 0, 4, 16, 28, 40 and 52 plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 299 | 294 | 289
Score on a scale | -11.7 [-12.3 to -11.1] | -11.2 [-11.8 to -10.5] | -9.5 [-10.1 to -8.9]
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, cLDA; [statistical method as in outcome 20, analysis 1]; Difference in least squares means = -1.7, 95% CI 2-sided [-2.4 to -1.0]
Statistical Analysis 2: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, cLDA; [statistical method as in outcome 20, analysis 1]; Difference in least squares means = -2.2, 95% CI 2-sided [-2.9 to -1.5]

22. Secondary Outcome: Change From Baseline in the DLQI at Week 40 (Part 3)
Description: The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Baseline and Week 40
Population: Participants who received at least one dose of study medication in Part 3 and with valid DLQI value at baseline and Week 40.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 108 | 107 | 212 | 58 | 21 | 21 | 69 | 65 | 114
Score on a scale | -11.6 (6.61) | -12.0 (7.11) | -13.2 (6.92) | -9.7 (5.62) | -9.0 (7.76) | -9.8 (7.25) | -10.4 (6.66) | -10.1 (6.08) | -10.8 (6.81)

23. Secondary Outcome: Change From Baseline in the DLQI at Week 52 (Part 3)
Description: as for outcome 22
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study medication in Part 3 and with valid DLQI value at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 104 | 205 | 58 | 19 | 19 | 65 | 63 | 114
Score on a scale | -11.3 (6.16) | -11.5 (7.26) | -13.1 (6.80) | -9.2 (6.18) | -9.4 (8.47) | -9.3 (7.22) | -11.1 (6.45) | -10.4 (6.38) | -11.5 (6.97)

24. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 12 (Part 1)
Description: as for outcome 19
Time Frame: Week 12
Population: Analysis population includes randomized participants who received at least one dose of study medication in Part 1 and with a valid DLQI value at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 306 | 296 | 150 | 304
Percentage of participants | 47.4 | 40.2 | 8.0 | 35.5
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 39.3, 95% CI 2-sided [31.8 to 46.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 32.1, 95% CI 2-sided [24.5 to 39.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Other; p = 0.003, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 11.9, 95% CI 2-sided [4.1 to 19.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Other; p = 0.221, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 4.8, 95% CI 2-sided [-2.9 to 12.5] — [estimate comment as in outcome 1, analysis 2]

25. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 28 (Part 2)
Description: as for outcome 19
Time Frame: Week 28
Population: Analysis population includes randomized participants to tildrakizumab 200 mg, tildrakizumab 100 mg or etanercept in Part 1, who received at least one dose of study medication in Part 2 and with a valid DLQI value at Week 28.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg
Number analyzed (Participants) | 297 | 290 | 282
Percentage of participants | 65.0 | 54.1 | 39.4
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 25.7, 95% CI 2-sided [17.7 to 33.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg vs Etanercept 50 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 15.0, 95% CI 2-sided [6.9 to 22.9] — [estimate comment as in outcome 1, analysis 2]

26. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 40 (Part 3)
Description: as for outcome 22
Time Frame: Week 40
Population: Participants who received at least one dose of study medication in Part 3 and with valid DLQI value at Week 40.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 108 | 108 | 212 | 60 | 21 | 21 | 69 | 66 | 116
Percentage of participants | 72.2 | 68.5 | 71.2 | 41.7 | 9.5 | 19.0 | 50.7 | 51.5 | 38.8

27. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 52 (Part 3)
Description: as for outcome 22
Time Frame: Week 52
Population: Participants who received at least one dose of study medication in Part 3 and with valid DLQI value at Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 105 | 105 | 205 | 60 | 19 | 19 | 65 | 64 | 116
Percentage of participants | 72.4 | 71.4 | 68.8 | 40.0 | 10.5 | 42.1 | 60.0 | 57.8 | 48.3

28. Secondary Outcome: Mean Change From Baseline in PASI Score Over Time (Part 1)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status.
Time Frame: Baseline and Week 4, Week 8 or Week 12
Population: Analysis population includes randomized participants who received at least one dose of study medication in Part 1 and with valid PASI value at baseline and at the time point for endpoint (ie, Weeks 4, 8 and 12).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 155 | 312
Scores on a scale
  Week 4: number analyzed (Participants) | 308 | 303 | 150 | 306
  Week 4 | -8.1 (6.54) | -7.9 (6.83) | -2.3 (6.18) | -7.0 (7.15)
  Week 8: number analyzed (Participants) | 302 | 299 | 146 | 298
  Week 8 | -13.1 (7.71) | -12.8 (7.57) | -3.1 (7.18) | -11.4 (8.77)
  Week 12: number analyzed (Participants) | 302 | 297 | 142 | 288
  Week 12 | -15.4 (7.77) | -15.1 (7.94) | -3.4 (6.77) | -13.5 (8.29)

29. Secondary Outcome: Mean Change From Baseline in PASI Score Over Time (Part 2)
Description: as for outcome 28
Time Frame: Baseline and Week 16, Week 22 or Week 28
Population: Analysis population includes randomized participants who received at least one dose of study medication in Part 2 and with valid PASI value at baseline and at the time point for endpoint (ie, Weeks 16, 22 and 28).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo (Part 1)/ Tildrakizumab 200 mg (Part 2): Participants received placebo to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 200 mg SC on Weeks 12 and 16 (Part 2) plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Placebo (Part 1)/ Tildrakizumab 100 mg (Part 2): Participants received placebo to tildrakizumab SC on Weeks 0 and 4 (Part 1), and tildrakizumab 100 mg SC on Weeks 12 and 16 (Part 2) plus etanercept placebo twice weekly until Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg | Placebo (Part 1)/ Tildrakizumab 200 mg (Part 2) | Placebo (Part 1)/ Tildrakizumab 100 mg (Part 2)
Number analyzed (Participants) | 314 | 307 | 312 | 72 | 68
Scores on a scale
  Week 16: number analyzed (Participants) | 298 | 291 | 283 | 72 | 68
  Week 16 | -16.2 (7.70) | -15.9 (7.87) | -14.2 (8.20) | -11.6 (6.97) | -9.6 (6.71)
  Week 22: number analyzed (Participants) | 293 | 290 | 281 | 71 | 67
  Week 22 | -17.1 (7.66) | -16.7 (7.88) | -14.5 (8.32) | -15.1 (6.55) | -13.7 (7.18)
  Week 28: number analyzed (Participants) | 293 | 290 | 277 | 68 | 66
  Week 28 | -17.0 (7.81) | -16.5 (7.71) | -14.8 (7.85) | -17.3 (7.62) | -14.5 (8.46)

30. Secondary Outcome: Mean Change From Baseline in PASI Score Over Time (Part 3)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. Week-28 responder (Wk-28 R) is a participant who achieved ≥ 75% improvement in PASI from baseline at Week 28. Week-28 partial responder (Wk-28 PR) is a participant who achieved ≥50% and <75% improvement in PASI response from baseline at Week 28.
Time Frame: Baseline and Week 32, Week 36, Week 40, Week 46 and Week 52
Population: Analysis population includes randomized participants who received at least one dose of study medication in Part 3 and with valid PASI value at baseline and at the time point for endpoint (ie, Weeks 32, 36, 40, 46 and 52).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 108 | 110 | 212 | 60 | 21 | 21 | 68 | 65 | 121
Scores on a scale
  Week 32: number analyzed (Participants) | 105 | 110 | 207 | 60 | 20 | 20 | 68 | 65 | 116
  Week 32 | -19.0 (7.13) | -19.0 (8.03) | -18.7 (6.83) | -14.0 (5.72) | -15.0 (6.69) | -15.5 (7.08) | -16.9 (7.68) | -16.4 (8.02) | -10.5 (6.25)
  Week 36: number analyzed (Participants) | 108 | 107 | 210 | 59 | 21 | 21 | 68 | 65 | 118
  Week 36 | -18.9 (7.11) | -19.0 (8.17) | -18.9 (7.18) | -14.5 (5.92) | -15.7 (8.09) | -16.0 (8.13) | -17.6 (6.80) | -16.7 (8.19) | -12.9 (6.64)
  Week 40: number analyzed (Participants) | 107 | 108 | 212 | 60 | 21 | 21 | 67 | 64 | 114
  Week 40 | -18.8 (7.04) | -18.5 (7.56) | -18.7 (6.95) | -14.4 (6.00) | -16.0 (8.73) | -16.5 (8.59) | -17.9 (7.03) | -16.9 (7.99) | -14.6 (6.42)
  Week 46: number analyzed (Participants) | 105 | 105 | 205 | 59 | 21 | 20 | 65 | 64 | 115
  Week 46 | -19.0 (7.13) | -18.1 (7.45) | -18.7 (6.76) | -14.5 (5.99) | -16.2 (8.76) | -15.8 (9.72) | -17.9 (6.24) | -17.1 (7.30) | -15.6 (7.16)
  Week 52: number analyzed (Participants) | 105 | 104 | 204 | 60 | 19 | 19 | 66 | 63 | 113
  Week 52 | -18.9 (7.13) | -18.4 (7.66) | -18.4 (6.65) | -14.6 (5.72) | -15.5 (9.00) | -16.3 (9.55) | -18.1 (7.00) | -17.0 (7.30) | -16.2 (6.83)

31. Secondary Outcome: Mean Percent Change From Baseline in PASI Score Over Time (Part 1)
Description: as for outcome 28
Time Frame: Baseline and Week 4, Week 8 or Week 12
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Placebo | Etanercept 50 mg
Number analyzed (Participants) | 314 | 307 | 155 | 312
Percent change
  Week 4: number analyzed (Participants) | 308 | 303 | 150 | 306
  Week 4 | -40.2 (27.86) | -39.3 (30.02) | -11.7 (30.37) | -33.9 (33.55)
  Week 8: number analyzed (Participants) | 302 | 299 | 146 | 298
  Week 8 | -65.7 (26.58) | -63.8 (29.65) | -15.3 (35.95) | -55.7 (35.10)
  Week 12: number analyzed (Participants) | 302 | 297 | 142 | 288
  Week 12 | -78.0 (22.31) | -74.8 (28.11) | -17.4 (32.95) | -66.7 (30.78)

32. Secondary Outcome: Mean Percent Change From Baseline in PASI Score Over Time (Part 2)
Description: as for outcome 28
Time Frame: Baseline and Week 16, Week 22 or Week 28
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tildrakizumab 200 mg | Tildrakizumab 100 mg | Etanercept 50 mg | Placebo (Part 1)/ Tildrakizumab 200 mg (Part 2) | Placebo (Part 1)/ Tildrakizumab 100 mg (Part 2)
Number analyzed (Participants) | 314 | 307 | 312 | 72 | 68
Percent change
  Week 16: number analyzed (Participants) | 298 | 291 | 283 | 72 | 68
  Week 16 | -82.0 (21.26) | -79.3 (25.27) | -70.3 (27.55) | -59.2 (28.34) | -49.4 (28.95)
  Week 22: number analyzed (Participants) | 293 | 290 | 281 | 71 | 67
  Week 22 | -86.6 (17.58) | -82.9 (23.16) | -71.9 (29.40) | -77.9 (20.25) | -70.1 (25.24)
  Week 28: number analyzed (Participants) | 293 | 290 | 277 | 68 | 66
  Week 28 | -85.7 (17.44) | -82.5 (22.33) | -73.5 (24.40) | -84.0 (16.89) | -72.9 (30.05)

33. Secondary Outcome: Mean Percent Change From Baseline in PASI Score Over Time (Part 3)
Description: as for outcome 30
Time Frame: Baseline and Week 32, Week 36, Week 40, Week 46 and Week 52
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1 & 2)/ 100 mg (Part 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 R | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) Wk-28 PR | Tildrakizumab 100 mg (Parts 1, 2, & 3) Wk-28 PR | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3) | Etanercept 50 mg (Parts 1 & 2)/ Tildrakizumab 200 mg (Part 3)
Number analyzed (Participants) | 108 | 110 | 212 | 60 | 21 | 21 | 68 | 65 | 121
Percent change
  Week 32: number analyzed (Participants) | 105 | 110 | 207 | 60 | 20 | 20 | 68 | 65 | 116
  Week 32 | -94.9 (6.19) | -94.0 (7.02) | -94.3 (7.33) | -77.1 (16.73) | -71.1 (13.21) | -75.3 (16.90) | -84.4 (24.18) | -81.6 (21.69) | -54.7 (24.05)
  Week 36: number analyzed (Participants) | 108 | 107 | 210 | 59 | 21 | 21 | 68 | 65 | 118
  Week 36 | -94.5 (7.47) | -94.0 (6.93) | -94.4 (7.06) | -79.9 (15.94) | -74.4 (15.69) | -77.9 (15.47) | -87.7 (15.20) | -83.1 (19.83) | -65.9 (21.35)
  Week 40: number analyzed (Participants) | 107 | 108 | 212 | 60 | 21 | 21 | 67 | 64 | 114
  Week 40 | -94.2 (7.69) | -92.6 (10.25) | -94.3 (7.40) | -79.1 (17.10) | -75.7 (19.24) | -80.6 (17.57) | -88.2 (14.55) | -84.1 (17.08) | -76.5 (17.98)
  Week 46: number analyzed (Participants) | 105 | 105 | 205 | 59 | 21 | 20 | 65 | 64 | 115
  Week 46 | -94.8 (7.77) | -91.4 (12.09) | -94.3 (7.64) | -79.3 (17.77) | -77.1 (19.67) | -75.3 (23.35) | -90.3 (12.32) | -86.9 (13.08) | -80.3 (17.92)
  Week 52: number analyzed (Participants) | 105 | 104 | 204 | 60 | 19 | 19 | 66 | 63 | 113
  Week 52 | -94.7 (8.06) | -92.2 (10.57) | -93.4 (9.81) | -80.4 (15.68) | -75.7 (36.00) | -79.6 (21.46) | -91.0 (12.16) | -87.1 (12.90) | -84.2 (16.07)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks (Part 1: Weeks 0-12; Part 2: Weeks 12-28; Part 3: Weeks 28-52)
Description: Part 1 includes all randomized participants who received at least 1 dose of Part 1 study drug, based on the treatment received. Part 2 includes all randomized participants who received at least 1 dose of Part 2 study drug, based on the treatment received, including those on placebo re-randomized at Week 12 to tildrakizumab. Part 3 includes all participants who received at least 1 dose of Part 3 study drug, based on the treatment received.
Groups:
- Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R: Participants received tildrakizumab 200 mg SC on Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28 and 40 (Part 3) plus etanercept PBO twice weekly until Week 12 and once weekly from Week 12 to Week 28.
- Tildrakizumab 100 mg (Parts 1, 2 & 3): Participants received tildrakizumab 100 mg SC on Weeks 0, 4 and then every 12 weeks.
- Placebo (Part 1): Participants received matching placebo to tildrakizumab SC on Weeks 0 and 4.
- Etanercept 50 mg (Parts 1 & 2): Participants received etanercept 50 mg twice weekly up to Week 12 and once weekly from Week 12 to Week 28.
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R | Tildrakizumab 100 mg (Parts 1, 2 & 3) | Placebo (Part 1) | Etanercept 50 mg (Parts 1 & 2)
All-Cause Mortality (participants affected / at risk) | 0/527 | 3/487 | 0/156 | 0/313
Serious Adverse Events (participants affected / at risk) | 26/527 | 30/487 | 4/156 | 20/313
Other Adverse Events (participants affected / at risk) | 167/527 | 151/487 | 23/156 | 118/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R (N=527) | Tildrakizumab 100 mg (Parts 1, 2 & 3) (N=487) | Placebo (Part 1) (N=156) | Etanercept 50 mg (Parts 1 & 2) (N=313)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy alcoholic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breact cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab 200 mg (Parts 1, 2 & 3) Wk-28 R (N=527) | Tildrakizumab 100 mg (Parts 1, 2 & 3) (N=487) | Placebo (Part 1) (N=156) | Etanercept 50 mg (Parts 1 & 2) (N=313)
Injection site erythema (General disorders) | 5 (7) | 5 (5) | 1 (2) | 28 (98)
Injection site reaction (General disorders) | 4 (8) | 2 (2) | 1 (1) | 17 (54)
Nasopharyngitis (Infections and infestations) | 119 (173) | 112 (152) | 12 (14) | 63 (79)
Upper respiratory tract infection (Infections and infestations) | 27 (30) | 15 (18) | 1 (1) | 11 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17) | 26 (30) | 3 (3) | 10 (13)
Headache (Nervous system disorders) | 30 (40) | 29 (46) | 6 (6) | 18 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the Sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.